CLINICAL TRIAL: NCT02914067
Title: Cognitive Biomarkers in Pediatric Brain Tumor Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Children's Discovery Institute (Other); Neurosurgery Research & Education Foundation (Unknown); The Andrew McDonough B+ Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201609023
Record Dates: First submitted 2016-09-19; First posted 2016-09-26 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Childhood Brain Tumor
Keywords: Pediatric brain tumors; Cognitive deficits; Resting state functional connectivity; NIH toolbox
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Cohort 1 (Experimental): * Prior to surgery, subjects will have a complete standard of care history and physical exam by the neurosurgeon and then undergo peri-diagnostic neurocognitive testing utilizing the NIH Toolbox Cognitive Battery computer testing software for iPad (will take 45 minutes). The peri-diagnostic period will be defined as the period from first presentation to 2 weeks post-diagnosis or two weeks post-op, whichever is later.
  * Participants will also undergo a rsfcMRI during their standard of care MRI imaging which will add 15 minutes to their scan time
  Interventions: Other: Neurocognitive testing; Device: rsfcMRI
- Cohort 2 (Experimental): * Patients with diagnosis of a posterior tumor will undergo neurocognitive testing utilizing the NIH Toolbox. Testing will be every 6 months for children currently receiving therapy and annually for those that have completed all therapy for a total of 3 sessions. During standard of care MRI images, rsfcMRI imaging will be performed which will add 15 minutes of time. rsfcMRI will be obtained every 6 months for children currently receiving therapy and annually for those that have completed therapy for a total of 3 rsfcMRIs for each patient.
  * Patients in Cohort 1 will also be eligible to continue with the longitudinal assessment as just described. These participants will then undergo repeat neurocognitive testing using the NIH toolbox 6-9 months for an additional 3 testing sessions. rsfcMRI will be obtained during their follow-up imaging at 6-9 month intervals for a total of 3 additional rsfcMRIs (4 total scans).
  Interventions: Other: Neurocognitive testing; Device: rsfcMRI
- Cohort 3 (Experimental): * During standard of care MRI images, rsfcMRI imaging will be performed which will add 15 minutes of scan time.
  * rsfcMRI will be obtained annually for total of 3 rsfcMRIs for each patient.
  Interventions: Device: rsfcMRI
- Cohort 4 Arm A (Experimental): Undergo the following MRI images: RSFC MRI, T2/T1 MRI, and DTI.
  * Will complete cognitive testing using the NIH Toolbox Cognitive Battery
  * All patients will complete the Attention Deficit/Hyperactivity Disorder (ADHD) Rating Scale - 5 questionnaire. All patients will complete a self-reported assessment of neurological quality of life (QOL). Adult patients (age ≥ 18 years) will complete the adult version of the Quality of Life in Neurological Disorders (Neuro-QOL) Cognitive Function measure. All pediatric patients will complete the pediatric version of the Neuro-QOL Cognitive Function measure. For patients <18 years of age and for adult patients with parent present, parent/caregiver will complete the PROMIS® Parent Proxy for cognition. All adult patients will complete the Colorado Learning Difficulties Questionnaire (CLDQ). This questionnaire will be completed by parent/caregiver for patients < 18 years of age.
  Interventions: Other: Neurocognitive testing; Device: rsfcMRI
- Cohort 4 Arm B (Experimental): * During standard of care MRI images, rsfcMRI imaging will be performed which will add 15 minutes of scan time.
  * Will complete cognitive testing using the NIH Toolbox Cognitive Battery
  * All patients will complete the Attention Deficit/Hyperactivity Disorder (ADHD) Rating Scale - 5 questionnaire. All patients will complete a self-reported assessment of neurological quality of life (QOL). Adult patients (age ≥ 18 years) will complete the adult version of the Quality of Life in Neurological Disorders (Neuro-QOL) Cognitive Function measure. All pediatric patients will complete the pediatric version of the Neuro-QOL Cognitive Function measure. For patients <18 years of age and for adult patients with parent present, parent/caregiver will complete the PROMIS® Parent Proxy for cognition. All adult patients will complete the Colorado Learning Difficulties Questionnaire (CLDQ). This questionnaire will be completed by parent/caregiver for patients < 18 years of age.
  Interventions: Other: Neurocognitive testing; Device: rsfcMRI

INTERVENTIONS:
Other: Neurocognitive testing
  Arms: Cohort 1; Cohort 2; Cohort 4 Arm A; Cohort 4 Arm B
Device: rsfcMRI — The imaging protocols will be a combined version of a standard of care (SOC) protocol with a research portion. The SOC portion of the pre-surgical scans includes a 3D T2-weighted (T2w) scans and 3D pre- and post-contrast T1-weighted (T1w) images, both at high resolution (1.0 mm3) for use in the intraoperative navigation system. This scan also includes a DTI portion for definition of fiber bundles of interest. The SOC portion of the post-surgical scans includes transverse FLAIR and post-contrast T1w images in all 3 planes. The research portion of the scan will be identical at all 3 time points and include 15 min of rsfcMRI during which the non-sedated subjects will be asked to stay still and awake while looking at a fixation cross

SUMMARY:
The investigators will focus on three cohorts of brain tumor patients aged, 4-18 years, to answer two critical questions: 1) Can the investigators acquire high quality data relevant to cognitive function during the peri-diagnostic period and, 2) can the investigators develop predictive models for cognitive outcomes using serial examination of functional imaging and cognitive function. Any patient with a newly diagnosed brain tumor aged 4-18 will be eligible for enrollment in cohort 1. Only patients with previously diagnosed tumors of the posterior fossa will be eligible for cohort 2. For cohort 3, eligible patients will include patients with a clinical diagnosis of posterior fossa syndrome with physical impairments that prohibit completion of the NIH Toolbox Cognitive Battery. The investigators have decided to expand the eligible tumor types to better capture the most significant deficit variability that can be caused by tumors outside the posterior fossa. Thus, this focus will provide a platform to analyze the impact that different tumor types and different standard treatments have on cognitive dysfunction. The rationale for inclusion of subjects on cohort 3 is that posterior fossa syndrome is one of the most cognitively devastating diagnoses following a posterior fossa surgery. The causes of posterior fossa syndrome and unknown and there are currently no interventions to improve symptoms. RsfcMRI would offer a novel and non-invasive assessment of posterior fossa syndrome patients by assessing connectivity within and outside of the cerebellum. Expanding the tumor eligibility will allow us to further explore the effect tumor location will have on cognitive testing and rsfcMRI. Here, repeated evaluations on and off therapy will provide the necessary data points to establish trajectories of cognitive development and recovery in this population.

ELIGIBILITY:
Cohort 1 (30 patients will be enrolled to this cohort)

Inclusion Criteria:

* Between 4 and 18 years of age, inclusive
* Newly diagnosed primary brain tumor of any location and any histology
* Life expectancy of at least one year
* Able to understand and willing to consent or assent to the research proposed, along with consent of legal guardian(s) if applicable

Exclusion Criteria:

* Presence of visual impairment to an extent that the patient is unable to complete the computer testing
* Contraindication to MRI scan (i.e. due to cardiac pacemaker)
* Programmable Shunt

Cohort 2 (150 patients will enrolled to this cohort. This may include some or all of the patients enrolled to Cohort 1.)

Inclusion Criteria:

* Between 4 and 18 years of age, inclusive
* Previous diagnosis of a posterior fossa brain tumor; patients who are either undergoing active treatment for posterior fossa tumor or who have completed treatment will be eligible for study enrollment
* Life expectancy of at least one year
* Able to understand and willing to consent assent to the research proposed, along with consent of legal guardian(s) if applicable

Exclusion Criteria:

* Presence of visual impairment to an extent that the patient is unable to complete the computer testing
* Contraindication to MRI scan (i.e. due to cardiac pacemaker)

Cohort 3 (20 patients will be enrolled to this cohort. This may include some or all of the patients enrolled to Cohort 1) Inclusion Criteria

* Between 4 and 18 years of age, inclusive
* Previous diagnosis of a posterior fossa brain tumor
* Clinical diagnosis of post-operative posterior fossa syndrome
* Inability to complete NIH Toolbox
* Life expectancy of at least one year
* Able to understand and willing to consent assent to the research proposed, along with consent of legal guardian(s) if applicable

Exclusion Criteria

* Contraindication to MRI scan (i.e. due to cardiac pacemaker)

Cohort 4 (50 Patients will be enrolled to Cohort 4. This will include patients previously enrolled on Cohorts 1-3 above.)

Inclusion Criteria

* Between 12-30 years of age, inclusive
* Diagnosis of a brain tumor >3 years prior to study enrollment
* Life expectancy of at least one year
* Able to understand and willing to consent assent to the research proposed, along with consent of legal guardian(s) if applicable
* Patient must be able to complete a 1 hour MRI scan without sedation

Exclusion Criteria

* Contraindiciation to MRI scan (i.e. due to cardian pacemaker)
* Presence of dental braces or programmable shunt
* Patient requires sedation for MRI scan

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-10-26 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Identify reliable peri-diagnostic estimators of cognition as measured by neurocognitive testing | Peri-diagnostic period (from first presentation to 2 weeks post-diagnosis or two weeks post-op, whichever is later)
Identify reliable peri-diagnostic estimators of cognition as measured by advanced resting-state functional connectivity MRI (rsfcMRI) data | Peri-diagnostic period (from first presentation to 2 weeks post-diagnosis or two weeks post-op, whichever is later)
Predictors of cognitive recovery in children as determined by multiplexed analyses of a combination of potential biomarkers across multiple modalities (rsfcMRI, structural MRI, NIH Toolbox, patient demographics, treatment information) | Up to 27 months
  As dictated by information theory, properly combining predictors across modalities must increase the accuracy of the prediction algorithm, unless a given modality contains no information about the question of interest (in this case, long-term cognitive outcomes).
Identify reliable peri-diagnostic estimators of brain function as measured by neurocognitive testing | Peri-diagnostic period (from first presentation to 2 weeks post-diagnosis or two weeks post-op, whichever is later)
Identify reliable peri-diagnostic estimators of brain function as measured by advanced resting-state functional connectivity MRI (rsfcMRI) data | Peri-diagnostic period (from first presentation to 2 weeks post-diagnosis or two weeks post-op, whichever is later)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Perkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu